CLINICAL TRIAL: NCT01229423
Title: Safety and Efficacy of LATISSE® in the Augmentation of Eyelashes of Korean Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAT-KOR-01
Record Dates: First submitted 2010-10-25; First posted 2010-10-27 (Estimated); Results first posted 2012-01-23 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Eyelash Hypotrichosis
MeSH Terms: interventions — Bimatoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LATISSE® (Experimental): bimatoprost 0.03% (LATISSE®)
  Interventions: Drug: bimatoprost 0.03%

INTERVENTIONS:
Drug: bimatoprost 0.03% — One drop of bimatoprost 0.03% (LATISSE®) applied evenly to each upper eyelid in the evening. Treatment is once daily for up to 40 weeks.
  Other Names: LATISSE®

SUMMARY:
This study will evaluate the safety and efficacy of LATISSE® (bimatoprost 0.03%) in the augmentation of eyelashes in Korean women.

ELIGIBILITY:
Inclusion Criteria:

* Eyelash prominence assessment of minimal or moderate
* Of Korean ethnicity

Exclusion Criteria:

* Any eye disease or abnormality
* Any ocular surgery or use of any eyelash extension or eyelash growth products within 3 months
* Any permanent eyeliner within 5 years
* Eyelash implants of any kind
* Eyelash tint or dye application within 2 months
* Use of any treatment that may affect hair growth within 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-11; Primary Completion 2010-06 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Seoul, South Korea

REFERENCES:
- [Background] Kwon O, Kim JY, Paik SH, Jeon HC, Jung YJ, Lee Y, Baek JH, Chun JH, Lee WS, Lee JY, Rogers JD, Halstead M, Eun HC. Long-term utility and durability of the therapeutic effects of bimatoprost 0.03% for eyelash augmentation in healthy Asian subjects. Dermatology. 2014;229(3):222-9. doi: 10.1159/000363379. Epub 2014 Sep 6. PMID 25228046

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LATISSE®
Started | 62
Completed | 47
Not Completed | 15

BASELINE CHARACTERISTICS:
Arm/Group | LATISSE®
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (6.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Eyelash Length at Week 20
Description: Change from baseline in eyelash length at Week 20. Measurements made were based on the mean length of the upper left and right eyelashes. A positive change from baseline indicates an increase in eyelash length, and a negative change from baseline indicates a decrease in eyelash length.
Time Frame: Baseline, Week 20
Population: Intent-to-Treat (ITT) included all patients enrolled in the trial who received at least one application of study drug.
Measure: Mean (Standard Deviation); unit: Millimeter (mm)
Arm/Group | LATISSE®
Number analyzed (Participants) | 62
Millimeter (mm)
  Baseline | 5.92 (0.72)
  Change from Baseline at Week 20 | 1.10 (0.8)

2. Secondary Outcome: Percentage of Subjects With an Improvement of at Least 1-Point in Global Eyelash Assessment (GEA) Score at Week 20
Description: Percentage of subjects with an improvement of at least 1-point in GEA score at Week 20 from baseline. The GEA scale is an investigator-graded 4-point scale of overall eyelash prominence where 1=minimal, 2=moderate, 3=marked, and 4=very marked prominence.
Time Frame: Week 20
Population: Intent-to-Treat (ITT) included all patients enrolled in the trial who received at least one application of study drug.
Measure: Number; unit: Percentage of Subjects
Arm/Group | LATISSE®
Number analyzed (Participants) | 62
Percentage of Subjects | 81.4

3. Secondary Outcome: Change From Baseline in Eyelash Thickness at Week 20
Description: Change from baseline in eyelash thickness at Week 20. Assessments made were based on the mean thickness of the upper left and right eyelashes. A positive change from baseline indicates an increase in eyelash thickness, and a negative change from baseline indicates a decrease in eyelash thickness.
Time Frame: Baseline, Week 20
Population: Intent-to-Treat (ITT) included all patients enrolled in the trial who received at least one application of study drug.
Measure: Mean (Standard Deviation); unit: Millimeters Squared (mm^2)
Arm/Group | LATISSE®
Number analyzed (Participants) | 62
Millimeters Squared (mm^2)
  Baseline | 1.39 (0.395)
  Change from Baseline at Week 20 | 0.25 (0.269)

4. Secondary Outcome: Change From Baseline in Eyelash Intensity (Darkness) at Week 20
Description: Change from baseline in eyelash intensity (darkness) at Week 20. Assessments made were based on the mean eyelash intensity of the upper left and right eyelashes. Intensity was measured on a scale ranging from 0 (black) to 255 (white). A negative change from baseline indicates eyelash darkening in color, and a positive change from baseline indicates eyelash lightening in color.
Time Frame: Baseline, Week 20
Population: Intent-to-Treat (ITT) included all patients enrolled in the trial who received at least one application of study drug.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | LATISSE®
Number analyzed (Participants) | 62
Units on a Scale
  Baseline | 140.02 (15.788)
  Change from Baseline at Week 20 | -12.97 (13.115)

5. Secondary Outcome: Percentage of Subjects With an Improvement in Satisfaction With Overall Eyelash Prominence at Week 20
Description: Percentage of subjects with an improvement in satisfaction with overall eyelash prominence at Week 20. Subject satisfaction with overall eyelash prominence was assessed by response to the question "Overall how satisfied are you with your eyelashes?" Responses were based on a 5-point scale ("very unsatisfied", "unsatisfied", "neutral", "satisfied", "very satisfied"). Improvement in subject satisfaction is defined as a 1-point increase from baseline.
Time Frame: Week 20
Population: Intent-to-Treat (ITT) included all patients enrolled in the trial who received at least one application of study drug.
Measure: Number; unit: Percentage of Subjects
Arm/Group | LATISSE®
Number analyzed (Participants) | 62
Percentage of Subjects | 83.05

6. Secondary Outcome: Percentage of Subjects Satisfied With Treatment at Week 20
Description: Percentage of subjects satisfied with treatment at week 20 was assessed using the Treatment Satisfaction Scale response to the question "Which best describes your satisfaction with LATISSE®?" Responses were "very satisfied", "satisfied", "neutral", "unsatisfied", and "very unsatisfied." Satisfied is defined as responses of "very satisfied" and "satisfied."
Time Frame: Week 20
Population: Intent-to-Treat (ITT) included all patients enrolled in the trial who received at least one application of study drug.
Measure: Number; unit: Percentage of Subjects
Arm/Group | LATISSE®
Number analyzed (Participants) | 62
Percentage of Subjects | 83.1

ADVERSE EVENTS:
Arm/Group | LATISSE®
Serious Adverse Events (participants affected / at risk) | 0/62
Other Adverse Events (participants affected / at risk) | 27/62
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LATISSE® (N=62)
Conjunctival Hyperaemia (Eye disorders) | 6
Nasopharyngitis (Infections and infestations) | 9
Hypertrichosis (Skin and subcutaneous tissue disorders) | 4
Skin Hyperpigmentation (eyelid) (Skin and subcutaneous tissue disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No